CLINICAL TRIAL: NCT07319806
Title: The Effect of Two Different Interventions on Emotional State, Pain, and Fear During Respiratory Panel Removal in Children: A Randomized Controlled Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Özge Karakaya Suzan, Asistant Doctor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: palm stimulator
Record Dates: First submitted 2025-12-20; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Procedural Pain; Fear Anxiety; Children
Keywords: Procedural Pain; Fear and Anxiety in Children; Palm Stimulator; Stress Ball; Emotional Behavior; Distraction Techniques; Pediatric Nursing
MeSH Terms: conditions — Pain, Procedural

STUDY DESIGN:
Intervention Model Description: This study uses a parallel-group randomized design in which eligible participants are assigned to one of three study arms: palm stimulator intervention, stress ball intervention, or routine care (control). Each participant receives only one intervention during the respiratory panel collection procedure and does not cross over to another group throughout the study period.
Who Masked: Outcomes Assessor
Masking Description: Only the outcome assessors responsible for scoring the observational measures and analyzing the study data are blinded to group allocation. Participants, caregivers, and the nurse delivering the intervention are not masked due to the visible nature of the non-pharmacological interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Palm Stimulator Intervention (Experimental): Participants in this arm will hold a palm stimulator device in their hand during the respiratory panel specimen collection procedure. The device provides tactile stimulation through surface protrusions designed to activate sensory input. The palm stimulator will be used only during the procedure and removed immediately after completion.
  Interventions: Behavioral: Palm Stimulator
- Stress Ball Intervention (Experimental): Participants in this arm will be provided with a stress ball during the respiratory panel specimen collection procedure. Children will be instructed to squeeze and release the stress ball repeatedly throughout the procedure as a distraction technique. The stress ball will be used only during the procedure.
  Interventions: Behavioral: Stress Ball
- Routine Care Control Group (No Intervention): Participants in this arm will receive routine care during the respiratory panel specimen collection procedure without the use of any additional non-pharmacological intervention. Standard clinical practices, including caregiver presence and verbal reassurance, will be applied.

INTERVENTIONS:
Behavioral: Palm Stimulator — Children will be instructed to hold the palm stimulator in the palm of their hand during the respiratory panel specimen collection procedure and to squeeze/grip it throughout the procedure as a tactile distraction strategy. The palm stimulator will be used only during the procedure and removed immediately after completion.
  Arms: Palm Stimulator Intervention
Behavioral: Stress Ball — Children will be given a stress ball during the respiratory panel specimen collection procedure and will be instructed to repeatedly squeeze and release the ball throughout the procedure as an active distraction technique (e.g., counting while squeezing). The stress ball will be used only during the procedure.
  Arms: Stress Ball Intervention

SUMMARY:
Respiratory panel collection is a commonly used diagnostic procedure in children with suspected respiratory tract infections; however, it is often perceived as painful and distressing. Inadequately managed pain and fear during such procedures may negatively affect children's emotional responses to future medical interventions.

This randomized controlled trial aims to evaluate and compare the effects of two non-pharmacological interventions-a palm stimulator and a stress ball-on pain, fear, and emotional behavior in children aged 6-12 years undergoing respiratory panel specimen collection. Participants will be randomly assigned to one of three groups: palm stimulator intervention, stress ball intervention, or routine care (control group).

Pain, fear, and emotional responses will be assessed using validated pediatric measurement tools before, during, and after the procedure. The findings of this study are expected to contribute evidence on simple, practical, and developmentally appropriate non-pharmacological strategies that can be safely integrated into pediatric nursing practice to improve children's procedural experiences.

DETAILED DESCRIPTION:
Procedural pain and fear are common challenges in pediatric clinical settings, particularly during invasive diagnostic procedures such as respiratory panel specimen collection. Children's negative emotional and behavioral responses during such procedures may lead to heightened distress, increased procedural resistance, and long-term fear of medical interventions. Therefore, the implementation of effective, safe, and developmentally appropriate non-pharmacological interventions is a priority in pediatric care.

This randomized controlled trial is designed to examine the comparative effectiveness of two tactile-based non-pharmacological interventions-a palm stimulator and a stress ball-on pain intensity, fear levels, and emotional behavior in children aged 6 to 12 years undergoing respiratory panel collection. The study adopts a parallel-group design with three arms: palm stimulator intervention, stress ball intervention, and routine care as the control condition.

Participants who meet the eligibility criteria will be randomly allocated to one of the three groups using a computer-generated randomization process. All respiratory panel specimen collections will be performed by the same trained pediatric nurse to minimize procedural variability. The interventions will be applied only during the specimen collection procedure, without altering standard clinical practice.

Pain, fear, and emotional responses will be assessed using validated pediatric measurement tools. Emotional behavior will be evaluated through structured behavioral observation before and after the procedure, while pain and fear will be assessed shortly after completion of the specimen collection. Assessments will be conducted by healthcare professionals who are not involved in the intervention delivery to reduce assessment bias.

By comparing two simple, low-cost, and easily applicable interventions with routine care, this study aims to generate evidence that can inform pediatric nursing practice and support the integration of non-pharmacological pain and fear management strategies into routine clinical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 12 years
* Hospitalized children scheduled for respiratory panel specimen collection
* Ability to communicate verbally, understand instructions, and follow commands
* Children not receiving sedative, anticonvulsant, or analgesic medications at the time of the procedure
* Written informed consent obtained from a parent or legal guardian
* Assent obtained from the child
* Willingness of the child and parent/legal guardian to participate in the study

Exclusion Criteria:

* Children who do not consent or assent to participate
* Children requiring more than one attempt for respiratory panel specimen collection
* Presence of chronic, acute, or life-threatening medical conditions
* Children with cognitive or communication impairments that prevent reliable assessment
* Children with dependence on electronic or technological devices that may interfere with the intervention

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity During Respiratory Panel Collection | Within 5 minutes after completion of the respiratory panel specimen collection
  Pain intensity will be assessed using the Wong-Baker FACES Pain Rating Scale. Children will rate the maximum level of pain experienced during the respiratory panel specimen collection procedure shortly after completion of the procedure. Higher scores indicate greater pain intensity.
Fear Level During Respiratory Panel Collection | Within 5 minutes after completion of the respiratory panel specimen collection
  Fear level will be measured using the Children's Fear Scale (CFS). Children will self-report their level of fear related to the respiratory panel specimen collection immediately after the procedure. Higher scores reflect greater fear.
Emotional Behavioral Response During Respiratory Panel Collection | From 2-3 minutes before the procedure to 2-3 minutes after completion of the respiratory panel specimen collection
  Emotional behavioral responses will be evaluated using the Children's Emotional Manifestation Scale. Behavioral observations will be conducted by a blinded outcome assessor before and after the respiratory panel specimen collection. Higher total scores indicate more negative emotional and behavioral responses.

CONTACTS AND LOCATIONS:
Locations (1):
- Düzce University, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No